CLINICAL TRIAL: NCT04805749
Title: Efficacy of Visceral Osteopathic Approach to Relieve Recurring Digestive Symptoms in Subjects With Inflammatory Bowel Diseases (IBS)
Brief Title: Osteopathic Approach in Inflammatory Bowel Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ecole Professionnelle des Osteopathes du Quebec (Other)
Responsible Party: Principal Investigator, Valérie Conway, Osteopath and Naturopath at Clinique Expertise Santé, PhD in food sciences, Ecole Professionnelle des Osteopathes du Quebec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSTEO in subjects with IBD
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Inflammatory Bowel Diseases (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Masking Description: The gut inflammation and gut permeability laboratory analysis will be performed by a independent laboratory testing services (FLUIDS iQ® Inc.,Ontario, Canada)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteopathic manipulation (Experimental): Spinal Mobilisation / Cranial Osteopathy therapy / Circulatory Techniques / Visceral osteopathic therapy
  Interventions: Other: Manual Therapy: osteopathy

INTERVENTIONS:
Other: Manual Therapy: osteopathy — Osteopathic protocol applied at week 0, 1, 2 and 3:
  1. Spinal mobilisation of L1, L2 and L3 vertebrae to stimulate the arterial supply of mesenteric attachments of the colon and small intestine.
  2. Visceral osteopathic therapy to address adhesions/ fixations in the presacral fascia, Toldt fascia, posterior peritoneum and caudal peritoneum.
  3. Circulatory techniques to stimulate the celiac plexus, the superior and inferior ganglia.
  4. Cranial osteopathy techniques to address the vagus parasympathetic nerves.

SUMMARY:
Crohn's disease (CD) and ulcerative colitis are bowel disease (IBS) with an autoimmune component believed to affect approximately 1 in 140 Canadians. Despite this high prevalence, more than 30% patients with IBD have to live with recurrent gastrointestinal symptoms that is poorly relieved by allopathic medicine. Numerous studies have shown that the quality of life of individuals with IBS is lower than that of the general population. Since visceral manipulations have been shown to be effective in reducing the main discomforts associated with IBS during clinical interventions, it seems likely that it may provide similar relief to patients with IBD. To our best knowledge, no study has evaluated the impact of osteopathic manual therapy on neuro-immuno-vascular modulation of intestine to reduce IBS symptoms.

The aim of this study is to assess the relevance of an osteopathic approach addressing the brain-intestine axis in order to improve symptomatology in subject suffering from IBD by modulating inflammation and vagal tone.

DETAILED DESCRIPTION:
For this study, 10 to 12 participant (18 to 65 years) with Inflammatory Bowel Disease (in remission state) will be recruited to receiving visceral osteopathic therapy. Participant will received four standardized osteopathic session of 45 minutes (1 session every 7 days: week 0, 1, 2 and 3) and a follow up visit at week 4. The osteopathic protocol will specifically address the gut-to-brain neuro-immuno-vascular axis.

Global quality of life and severity of IBS-like symptoms will be a assess at week 0, 2 and 4 using three standardized questionnaires. Gut permeability and intestinal inflammation will be assessed at week 0 and 4 by measuring Zonulin (pre-Haptoglobin 2), Histamine and Diamine Oxidase (DO) levels respectively. Vagal tone at the beginning and at the end of each osteopathic session will be evaluate using heart rate variability (HRV) measurements.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with inflammatory bowel disease (IBD) in remission state;
* Subjects must suffer form recurrent digestive symptoms fulfilling the Rome III criteria;
* Subjects' eating habits should be stable prior to the study.

Exclusion Criteria:

* Concomitant diagnosis of celiac disease or multiple food intolerance;
* Concomitant diagnosis of rheumatologic disease;
* Obesity (BMI ≥ 30);
* Concomitant diagnosis of severe depression or severe anxiety;
* Unstable thyroid or kidney condition;
* Subjects on antidepressant, anti-inflammatory (steroids) or analgesic (paracetamol, aspirin) will be excluded from the study;
* Smokers, patients with problematic alcohol consumption or consuming drugs will be excluded from the study;
* High performance athletes will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change from baseline in gut permeability marker | Week 0 (baseline); Week 4
  Zonulin (pre-Haptoglobin 2) on dried blood spot will be performed by FLUIDS iQ's analytical testing services (Intestinal iQ™ test kit).
  Zonulin (Pre-Haptoglobin 2) is a protein found in intestinal cells, with production and release mimicking the effect of certain bacterial toxins on the tight junctions of the small intestine. Zonulin binds to a specific receptor only on the luminal surface of the intestinal epithelia and triggers a cascade of biochemical processes that induces tight junction (TJ) disassembly and a subsequent permeability increase of the intestinal epithelia. The Zonulin range is from 1 to 20 ng/ml.
  Values between 1 and 6 ng/ml are considered as optimal Values between 6 and 10 ng/ml are considered as borderline Values from 10 to 20 ng/ml are considered as elevated
Mean Change from baseline in intestinal inflammation markers | Week 0 (baseline); Week 4
  Histamine (ng/ml), Diamine Oxidase (DAO) on dried blood spot will be performed by FLUIDS iQ's analytical testing services (Intestinal iQ™ test kit).
  HISTAMINE
  * Normal reference range: 0.2 to 2.4 ng/ml
  * Below reference range: < 0.2 ng/ml
  * Above reference range: > 2.4 ng/ml
  DAO
  * Normal reference range: 12.5 to 3.75 ng/ml
  * Below reference range, < 3.75 ng/ml
  * Above reference range, > 12.5 ng/ml
Mean Change from baseline in vagally mediated Heart Rate Variability (HRV) | Week 0 ; Week 1; Week 2; Week 3
  The root mean square of successive differences between normal heartbeats (RMSSD) and Heart Rate Variability (HRV) will be recorded using Ultra-Short-Term measurement protocol (1-min resting). HRV and RMSSD will be measured at the start and at the end of each session.
  *Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Frontiers in Public Health. 2017;5(258).

SECONDARY OUTCOMES:
Mean Change from baseline in Irritable Bowel Syndrome (IBS) like symptoms | Week 0 (baseline); Week 2; Week 4
  Irritable Bowel Severity Scoring System (IBS-SSS)*
  The maximum severity of symptom score achievable is 500
  * Normal score <75 (remission)
  * Mild score: 75-174
  * Moderate score:175-300
  * Severe score: >300
    * Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997;11(2):395-402.
Mean Change from baseline in Quality of Life Score | Week 0 (baseline); Week 2; Week 5
  Irritable Bowel Syndrome Quality Of Life assessment (IBS-QOL)*
  34 items (scale 1 to 5) consisting of 8 subscale domains. The maximum score achievable is 175
  Sub-scale domains:
  * Dysphoria: 8 items; maximum score = 40
  * Interference with activity: 7 items; maximum score = 35
  * Body image: 4 items; maximum score= 20
  * Health worry: 3 items; maximum score = 15
  * Food avoidance 3 items; maximum score = 15
  * Social reaction 4 items; maximum score = 20
  * Sexual: 2 items; maximum score = 10
  * Relationship: 3 items; maximum score = 15
    * Patrick DL, Drossman DA, Frederick IO, DiCesare J, Puder KL. Quality of life in persons with irritable bowel syndrome: development and validation of a new measure. Dig Dis Sci. 1998;43(2):400-11.
Mean Change from baseline in Anxiety and Depression Score | Week 0 (baseline); Week 4
  Anxiety and depression levels according to the Hospital Anxiety And Depression Scale questionnaire (HADS)*
  0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
  *Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003;1:29.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Conway, PhD, Principal Investigator — Clinique Expertise Santé

IPD SHARING:
Plan to Share IPD: No